CLINICAL TRIAL: NCT04112095
Title: Adherence With Continuous-dose Oral Contraceptive: Evaluation of Self-Selection and Use (ACCESS)
Brief Title: Adherence With Continuous-dose Oral Contraceptive: Evaluation of Self-Selection and Use
Acronym: ACCESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 151042-004
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Contraception
Keywords: Daily birth control
MeSH Terms: interventions — Norgestrel

STUDY DESIGN:
Intervention Model Description: Drug: Norgestrel 0.075 mg tablets All subjects enrolled in the use phase of this open-label study will be given the opportunity to purchase and take one Norgestrel 0.075 mg tablet daily up to 24 weeks.
  Subjects will use the investigational product based on their understanding of the directions on the outer packaging called the Drug Facts Label and information inside the product packaging called the Consumer Information Leaflet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Use Phase Norgestrel 0.075 mg (Experimental): Norgestrel 0.075 mg tablets to be taken orally, one tablet daily at the same time every day for up to 24 weeks
  Interventions: Drug: Norgestrel 0.075 mg tablets

INTERVENTIONS:
Drug: Norgestrel 0.075 mg tablets — All subjects enrolled in the use phase of this open-label study will be given the opportunity to purchase and take one Norgestrel 0.075 mg tablet daily up to 24 weeks.
  Subjects will use the investigational product based on their understanding of the directions on the outer packaging called the Drug Facts Label and information inside the product packaging called the Consumer Information Leaflet.

SUMMARY:
This study is designed to assess whether consumers select and use norgestrel 0.075 mg, a progestin only pill for contraception, in a manner consistent with the OTC package directions in an Over-the-Counter (OTC)-like setting.

DETAILED DESCRIPTION:
Subjects will be primarily recruited via passive recruiting methods, such as in-store posters, direct mail postcards, and digital space advertising.

Respondents to advertisements will either call the study phone line or visit the study website for prescreening and scheduling of an in-person enrollment visit at a local participating research site.

During the face-to-face enrollment visit, potential subjects who meet the inclusion and exclusion criteria for the study will be given an (empty) study medication package and will be allowed as much time as they need to review the information on the outside of the entire package. Subjects will then be asked if the product is OK or not OK for them to use.

Qualified subjects then will be allowed to obtain (pharmacy sites) or be given (clinic sites) the study product.

Approximately 35 sites will be used, comprising retail pharmacy research sites and women's health clinics or adolescents' clinics.

ELIGIBILITY:
Inclusion Criteria:

* Women who are willing to purchase (in the pharmacies) or be provided (in the clinics, for women younger than 18 years old) oral contraception for their own use for the purposes of the study

Exclusion Criteria:

* Cannot read, speak and understand English
* Cannot see well enough to read information on the label

Min Age: 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 962 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Self-Selection: Proportion of self-selection population who make a correct selection decision regarding use of the product. | One Day
  Measurement tool: interview
Actual Use: Proportion of Active Use Study Days on which a subject reported taking the product. | Up to 24 Weeks
  Measurement tool: electronic diary
Actual Use: Proportion of subjects who are adherent to daily dosing instructions. | Up to 24 Weeks
  Measurement tool: electronic diary
Actual Use: Proportion of Active Use Study Days on which a subject reported taking the product at the same time of the day. | Up to 24 Weeks
  Measurement tool: electronic diary

SECONDARY OUTCOMES:
Self-Selection: Proportion of self-selection population who are inappropriate for use who make a correct decision regarding non-selection of the product. | One Day
  Measurement tool: interview
Actual Use: Proportion of Active Use Study Days on which a subject reported taking the product, accounting for appropriate mitigating behaviors. | Up to 24 Weeks
  Measurement tool: electronic diary
Actual Use: Proportion of subjects who are adherent to daily dosing instructions, accounting for appropriate mitigating behaviors. | Up to 24 Weeks
  Measurement tool: electronic diary
Actual Use: Proportion of Active Use Study Days on which a subject reported taking the product within 27 hours of the previous dose, accounting for appropriate mitigating behaviors. | Up to 24 Weeks
  Measurement tool: electronic diary
Actual Use: Actual Use: Proportion of packs transitions without any missed pills between packs. | Up to 24 Weeks
  Measurement tool: electronic diary
Actual Use: Proportion of user population who do not use study medication together with another form of hormone containing birth control. | Up to 24 Weeks
  Measurement tool: phone interview and electronic diary
Actual Use: Proportion of user population who report using a barrier method of contraception (or abstaining from intercourse) for the first 48 hours after starting to use the study medication. | Two Days
  Measurement tool: electronic diary
Self-Select/Use: Proportion of self-select population taking products listed in the "ask a doctor or pharmacist before use" section of the label who do not select, who select but do not use, or who report contacting a HCP on product use. | Up to 24 Weeks
  Measurement tool: phone interview
Actual Use: Proportion of user population who become pregnant during the course of the study who report stopping use and seeking healthcare as directed by the label. | Up to 24 Weeks
  Measurement tool: phone interview
Actual Use: Proportion of user population who develop sudden or severe pain in their lower belly during the course of the study who report seeking healthcare as directed by the label. | Up to 24 Weeks
  Measurement tool: phone interview
Use: Proportion of users having a late period after missing any pills in the last month, not having a period for 2 months during the course of the study who report doing a pregnancy test or seeking healthcare as directed by the label or who stop use. | Up to 24 Weeks
  Measurement tool: phone interview
Actual Use: Proportion of user population who experience periods that last more than 8 days or are unusually heavy during the course of the study who report seeking healthcare as directed by the label or who stop use. | Up to 24 Weeks
  Measurement tool: phone interview
Actual Use: Proportion of user population who experience repeated vaginal bleeding brought on by sex during the course of the study who report seeking healthcare as directed by the label or who stop use. | Up to 24 Weeks
  Measurement tool: phone interview
Actual Use: Proportion of user population who start having migraines with aura or whose migraines get worse during the course of the study who report seeking healthcare as directed by the label or who stop use. | Up to 24 Weeks
  Measurement tool: phone interview
Actual Use: Proportion of user population who develop yellowing of the skin or whites of the eyes during the course of the study who report seeking healthcare as directed by the label. | Up to 24 Weeks
  Measurement tool: phone interview
Actual Use: Number of pregnancies reported during the course of the study that occur while taking the product. | Up to 24 Weeks
  Measurement tool: phone interview

CONTACTS AND LOCATIONS:
Overall Officials: Russ Bradford, MD, MSPH, Principal Investigator — Pegus Research, Inc.
Locations (38):
- United States (38):
  - HRA Pharma Investigational site 1012, Birmingham, Alabama
  - HRA Pharma Investigational Site 1008, Homewood, Alabama
  - HRA Pharma Investigational Site 1038, Mesa, Arizona
  - HRA Pharma Investigational Site 1032, Phoenix, Arizona
  - HRA Pharma Investigational Site 1027, Cerritos, California
  - HRA Pharma Investigational Site 1039, Downey, California
  - HRA Pharma investigational site 1035, Long Beach, California
  - HRA Pharma Investigational Site 1017, Long Beach, California
  - HRA Pharma Investigational Site 1034, Los Angeles, California
  - HRA Pharma Investigational Site 1029, Los Angeles, California
  - HRA Pharma Investigational Site 1028, Los Angeles, California
  - HRA Pharma Investigational Site 1033, Aurora, Colorado
  - HRA Pharma Investigational Site 1023, Dalton, Georgia
  - HRA Pharma Investigational Site 1018, Griffin, Georgia
  - HRA Pharma Investigational Site 1014, Rosedale, Maryland
  - HRA Pharma Investigational Site 1019, Framingham, Massachusetts
  - HRA Pharma Investigational Site 1011, Andover, Minnesota
  - HRA Pharma Investigational Site 1006, Elk River, Minnesota
  - HRA Pharma Investigational Site 1003, Saint Francis, Minnesota
  - HRA Pharma Investigational Site 1020, Saint Louis Park, Minnesota
  - HRA Pharma Investigational Site 1009, Albuquerque, New Mexico
  - HRA Pharma Investigational Site 1007, Albuquerque, New Mexico
  - HRA Pharma Investigational Site 1030, Bronxville, New York
  - HRA Pharma Investigational Site 1013, New York, New York
  - HRA Pharma Investigational Site 1037, The Bronx, New York
  - HRA Pharma Investigational Site 1031, The Bronx, New York
  - HRA Pharma Investigational Site 1015, Burlington, North Carolina
  - HRA Pharma Investigational Site 1002, South Charleston, Ohio
  - HRA Pharma Investigational Site 1036, Lafayette Hill, Pennsylvania
  - HRA Pharma Investigational Site 1025, Philadelphia, Pennsylvania
  - HRA Pharma investigational site 1016, Clarksville, Tennessee
  - HRA Pharma Investigational Site 1022, Houston, Texas
  - HRA Pharma Investigational Site 1001, Houston, Texas
  - HRA Pharma investigational site 1024, Mapleton, Utah
  - HRA Pharma Investigational Site 1040, Salt Lake City, Utah
  - HRA Pharma Investigational Site 1021, Enumclaw, Washington
  - HRA Pharma Investigational site 1005, Seattle, Washington
  - HRA Pharma Investigational site 1010, Snohomish, Washington

IPD SHARING:
Plan to Share IPD: No